CLINICAL TRIAL: NCT07357714
Title: Longitudinal Study on Urinary Function and Multimorbidity Risks Among Beijing Community-dwelling Elderly UFMR-BCE Longitudinal Study
Brief Title: Urinary Function and Multimorbidity Risks: A Longitudinal Study in Beijing Community-Dwelling Elderly
Acronym: UFMR-BE
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qing Yuan, Associate Chief Physician, Chinese PLA General Hospital
Other Study IDs: UFMR-BE
Record Dates: First submitted 2025-12-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Overactive Bladder; Benign Prostatic Hyperplasia; Female Pelvic Floor Dysfunction; Lower Urinary Tract Symptoms; Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus
Keywords: Beijing community-dwelling elderly; Urinary function; Multimorbidity; Longitudinal study; Age-related functional decline
MeSH Terms: conditions — Renal Insufficiency, Chronic; Urinary Bladder, Overactive; Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 1. Blood samples: Including whole blood, serum, and plasma; retained for subsequent omics detection (genomics, proteomics, metabolomics) and analysis of biochemical/metabolic indicators related to urinary function and multimorbidity.
  2. Urine samples: Retained for urinary function assessment (e.g., urine composition analysis, urinary marker detection) and exploration of associations between urinary biomarkers and age-related urinary system diseases (e.g., Overactive Bladder, Benign Prostatic Hyperplasia).
  3. Fresh frozen tissue samples: Retained (when clinically available and with informed consent) for in-depth study of pathological mechanisms underlying urinary system diseases and multimorbidity interactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Beijing Community Elderly: This is a single observational cohort (no intervention applied) consisting of Beijing community-dwelling residents aged ≥60 years who meet the study's eligibility criteria (inclusion: able to cooperate with questionnaires; exclusion: severe mental illness, end-stage disease, or expected lifespan <1 year). The cohort is established to prospectively track changes in urinary function (e.g., indicators of chronic kidney disease, overactive bladder, benign prostatic hyperplasia) and the occurrence/progression of multimorbidity (e.g., metabolic syndrome, cardiovascular diseases, diabetes) over time. It serves to analyze the dynamic association between age-related urinary function decline and multimorbidity, without implementing any experimental treatments or interventions-only collecting natural health data, biological samples, and follow-up outcomes (e.g., functional decline, disease diagnosis, death) as part of routine observation.

SUMMARY:
This study focuses on Beijing community residents aged 60 and above, aiming to understand how urinary function (like bladder or kidney function) and multiple health problems (such as high blood pressure, diabetes) affect each other as people age-since current studies often only look at single diseases and don't cover this group well. To join, participants need to be a 60+ Beijing community resident who can answer simple questions; those with serious mental illnesses or expected lifespan under 1 year can't take part. The study starts with a baseline check (asking about the participants' health, habits, doing blood/urine tests or urinary function assessments, and possibly collecting small blood/urine samples). After that, the investigators will follow up every 6-12 months (via phone or clinic to update health info) and repeat key checks yearly; people with lower cognitive ability will be checked every 3 months. The investigators will also record new illnesses, mobility issues (like falls), or death. The study has passed ethical review-participants will get clear info before joining, can quit anytime, and participants' data will stay private; participants will also get free health check reports and basic advice. For participants, this means regular health monitoring; for everyone, it'll help make tools to spot high-risk groups (like a community app), design better help (e.g., exercise plans), and push for yearly urinary health checks in communities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Permanent resident of the participating Beijing community
* Able to cooperate with and complete study questionnaires and related procedures

Exclusion Criteria:

* Severe mental illness that impairs ability to cooperate with the study
* End-stage disease (confirmed by clinical diagnosis)
* Clinically assessed life expectancy < 1 year

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is derived from community-dwelling elderly residents in Beijing. Specifically, it includes individuals aged 60 years and older who live permanently in Beijing's communities (not in hospitals, nursing homes, or other institutional care settings) and are able to participate in routine health assessments and follow-ups. This population covers a broad age spectrum, ranging from young elderly (60-69 years) to super-elderly (90 years and older), and reflects the general health and living characteristics of Beijing's community-residing elderly group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual Incidence of Age-Related Multimorbidity Associated with Urinary Function | Baseline (at enrollment), 12 months after enrollment (1st annual assessment), 24 months after enrollment (2nd annual assessment), through study completion (average follow-up duration: 3 years)
  This outcome measures the incidence of newly developed chronic multimorbidities closely linked to age-related urinary function changes, including metabolic syndrome, cardiovascular diseases, diabetes mellitus, and Alzheimer's disease. Diagnosis is confirmed by clinical diagnostic criteria (e.g., diabetes mellitus defined as fasting blood glucose ≥7.0 mmol/L; hypertension, a subtype of cardiovascular disease, defined as blood pressure ≥140/90 mmHg) combined with medical record review. It reflects the initial association between urinary function and systemic multimorbidity during the aging process. The unit of measurement is "incidence rate (%)".
Annual Progression Rate of Age-Related Multimorbidity Associated with Urinary Function | Baseline (at enrollment), 12 months after enrollment (1st annual assessment), 24 months after enrollment (2nd annual assessment), through study completion (average follow-up duration: 3 years)
  This outcome measures the proportion of participants with pre-existing multimorbidities (as specified above) who experience disease deterioration during follow-up. Progression is confirmed by clinical examinations and medical record review, including escalation of disease severity (e.g., progression from grade 1 to grade 2 hypertension) or occurrence of complications (e.g., diabetic nephropathy). It reflects the interactive worsening trend between urinary function and multimorbidity with aging. The unit of measurement is "progression rate (%)".
Annual Change in International Prostate Symptom Score (IPSS) | Baseline (at enrollment), 12 months after enrollment (1st annual follow-up), 24 months after enrollment (2nd annual follow-up), through study completion (average follow-up duration: 3 years)
  This outcome assesses the annual change in the severity of lower urinary tract symptoms (LUTS) using the standardized IPSS scale (range: 0-35 points). A higher score indicates more severe symptoms such as frequent urination, urgent urination, and dysuria. Participants complete the questionnaire under the guidance of trained healthcare professionals, and data are directly extracted from the scale results. It is a key indicator reflecting core urinary function symptoms. The unit of measurement is "change in score (points)".
Annual Change in Maximum Urinary Flow Rate (Qmax) | Baseline (at enrollment), 12 months after enrollment (1st annual follow-up), 24 months after enrollment (2nd annual follow-up), through study completion (average follow-up duration: 3 years)
  This outcome measures the annual change in the maximum speed of urination, which directly reflects bladder contractile function and urinary tract patency. Qmax is measured using a uroflowmeter, with participants required to empty their bladders completely during the test; the device automatically records the maximum flow rate. The unit of measurement is "change in value (mL/s)".
Annual Change in Post-Void Residual Urine Volume | Baseline (at enrollment), 12 months after enrollment (1st annual follow-up), 24 months after enrollment (2nd annual follow-up), through study completion (average follow-up duration: 3 years)
  This outcome assesses the annual change in the volume of urine remaining in the bladder after voiding, which reflects bladder emptying function. The measurement is performed by professional physicians using ultrasound, and results are reported in milliliters (mL). A volume >50 mL indicates bladder emptying dysfunction. The unit of measurement is "change in volume (mL)".

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This study implements a data management plan centered on privacy protection and regulatory compliance. Individual Participant Data (IPD), including participants' demographic details, health indicators, and biological sample data, is collected via standardized forms and stored in encrypted databases with access controls (e.g., role-based permission management).
  IPD might not be shared primarily due to privacy protection requirements. IPD contains sensitive personal health information, which is strictly regulated by laws such as the Personal Information Protection Law and ethical review commitments. Sharing IPD would require explicit informed consent from each participant, and unauthorized sharing risks privacy leakage (e.g., medical history exposure leading to discrimination). Given the sensitivity of elderly participants' health data, non-sharing is adopted to avoid potential harms and ensure compliance.